CLINICAL TRIAL: NCT05873946
Title: Evaluating the Impact of 2D Non-Navigated Intraoperative Ultrasound on Extent of Resection and Patients' Outcome in Glioma Surgery: A Retrospective Study
Brief Title: Assessing the Effectiveness of 2D Non-Navigated Intraoperative Ultrasound in Glioma Surgery
Acronym: 2D-ioUS-Glio
Status: Completed | Type: Observational
Sponsor: Hospital del Rio Hortega (Other)
Responsible Party: Principal Investigator, Santiago Cepeda, Principal Investigator, Hospital del Rio Hortega
Other Study IDs: 21-PI085-B
Record Dates: First submitted 2023-05-16; First posted 2023-05-24 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Glioma; Glioma, Malignant; Low-grade Glioma; High-grade Glioma; Glioblastoma
Keywords: Glioma; Low-grade glioma; High-grade glioma; intraoperative ultrasound; extent of resection
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Operated gliomas: Patients consecutively operated with a pathological diagnosis of glial tumor
  Interventions: Diagnostic Test: intraoperative ultrasound

INTERVENTIONS:
Diagnostic Test: intraoperative ultrasound — Use of 2D non-navigated intraoperative ultrasound as an operative adjunct

SUMMARY:
This retrospective study aims to assess the utility of 2D non-navigated intraoperative ultrasound (ioUS) as a cost-effective alternative for guiding the surgical resection of gliomas and for detecting residual tumor. The study will analyse the records from consecutive adult patients diagnosed with gliomas, undergoing craniotomy between June 2018 and June 2023. The extent of resection (EOR) will be determined using postoperative MRI as the gold standard. The study will also examine the sensitivity and specificity of ioUS in detecting residual tumor. This research seeks to determine if ioUS can be an affordable and reliable tool that, combined with other intraoperative adjuncts, may aid neurosurgeons in achieving the maximum safe resection in glioma surgery.

DETAILED DESCRIPTION:
Objective:

The objective of this retrospective study is to evaluate the effectiveness and utility of 2D non-navigated intraoperative ultrasound (ioUS) as a cost-effective method for guiding the surgical resection of gliomas and detecting residual tumor.

Methods:

The study will retrospectively analyze the records of consecutive adult patients diagnosed with gliomas who underwent craniotomy between June 2018 and June 2023. The patients' records must show that they underwent both intraoperative ultrasound and postoperative MRI.

Evaluation Criteria:

The primary evaluation metric will be the extent of resection (EOR), which will be determined using postoperative MRI scans as the gold standard. The EOR will be classified into gross total resection (GTR), near-total resection (NTR), subtotal resection (STR), and partial resection (PR) based on the MRI scans.

The study will also examine the sensitivity and specificity of ioUS in detecting residual tumor postoperatively. This analysis will help determine the accuracy of ioUS in predicting residual tumor that may not have been apparent during the surgical procedure.

Expected Outcomes:

The study aims to determine if ioUS can be a reliable and affordable tool for guiding the surgical resection of gliomas. If successful, ioUS, in conjunction with other intraoperative adjuncts, may provide a cost-effective method to aid neurosurgeons in achieving the maximum safe resection in glioma surgery.

The results of this study could have significant implications for the management of glioma patients, potentially leading to improved surgical outcomes, decreased postoperative complications, and ultimately, improved patient survival and quality of life.

The data collected from this retrospective analysis could also provide valuable insights for future prospective studies and could contribute to the development of guidelines for the use of ioUS in neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older.
* Patients diagnosed with gliomas, confirmed by a pathologist.
* Patients who are scheduled to undergo craniotomy for tumor resection.
* Patients who are willing and able to give informed consent for participation in the trial.
* Patients who are capable of undergoing both intraoperative ultrasound and postoperative MRI.

Exclusion Criteria:

* Patients under the age of 18.
* Patients with non-glioma brain tumors.
* Patients who underwent stereotactic biopsies.
* Patients who are unable to provide informed consent due to cognitive impairment, language barriers, or any other reason.
* Patients with contraindications for MRI such as certain types of implanted medical devices, severe claustrophobia, or allergies to contrast material.
* Pregnant or breastfeeding women.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population for this clinical trial will comprise of adult patients aged 18 years or older who have been diagnosed with gliomas. The population will likely reflect a diverse range of glioma types and stages, providing a comprehensive assessment of the effectiveness of the 2D non-navigated intraoperative ultrasound in the surgical management of these tumors.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Extent of tumor resection | 24 hours after the surgery
  Percentage of tumor removal

SECONDARY OUTCOMES:
Postoperative neurological deficit | From 24 hours to 30 days after the surgery
  Neurological deficit after the surgery determined by physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Cepeda, MD.,PhD., Principal Investigator — Department of Neurosurgery, Río Hortega University Hospital
Locations (1):
- University Hospital Rio Hortega, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cepeda S, Garcia-Garcia S, Arrese I, Sarabia R. Non-navigated 2D intraoperative ultrasound: An unsophisticated surgical tool to achieve high standards of care in glioma surgery. J Neurooncol. 2024 May;167(3):387-396. doi: 10.1007/s11060-024-04614-5. Epub 2024 Feb 28. PMID 38413458